CLINICAL TRIAL: NCT06610539
Title: A Prospective Open Label Study of Patient Reported Outcome Measures and Efficacy Following the Use of 1ml Magtrace® for Sentinel Lymph Node Biopsy in Breast Cancer Patients Undergoing Lumpectomy
Brief Title: PAS 1ml Magtrace® for Sentinel Lymph Node Biopsy in Breast Cancer Patients
Acronym: MAGProm
Status: Recruiting | Type: Observational
Sponsor: Endomagnetics Ltd. (Industry)
Collaborators: Endomagnetics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: US-004
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Magtrace; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to provide prospective evidence in the US population of the frequency of skin discoloration and Sentinel Lymph Node detection rate in patients who have recevied Magtrace for Sentinel Lymph Node Biopsy (SLNB) and to evaluate the impact that skin discoloration has on patients when it does occur using patient reported outcome measures.

DETAILED DESCRIPTION:
The purpose of this study is to provide prospective evidence in the US population of the frequency of skin discoloration and Sentinel Lymph Node (SLN) detection rate in patients who have received 1ml Magtrace for Sentinel Lymph Node Biopsy (SLNB) and to evaluate the impact that skin discoloration has on patients when it does occur using patient reported outcome measures utilising BREAST-Q.

Baseline assessment using BREAST-Q will performed. A key secondary objective is to demonstrate non-inferiority of sentinel lymph node (SLN) detection rate with Magtrace compared to the American Society of Breast Surgeons (ASBRS) performance standards.

All participants will undergo lymph node mapping with Magtrace, and Sentinel Lymph Node Biopsy undertaken and nodes localised with the Sentimag system, A sentimag count will be recorded for each node removed.

After completion of the surgery, at the postoperative visit the presence of Magtrace related discoloration will be assessed by the Investigator. Participants found to have no Magtrace related discoloration will be asked to complete the Post-Op BREAST-Q assessment and return at 12 months post-op for a follow-up visit. Those patients assessed as having the presence of Magtrace related skin discoloration will be asked complete the post-op BREAST-Q and will then undergo assessment of the size and severity of the discoloration. They will then be asked to return at 6, 12, 18 and 24 months for follow-up visits, or until the discoloration has resolved. At each of these visits the BREAST-Q will be completed, and the size and severity assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to give informed consent for participation in the study
* Patient is aged 18 years or older at the time of consent
* Patients undergoing planned breast conserving surgery (for example, lumpectomy or partial mastectomy) and SLNB with Magtrace

Exclusion Criteria:

* The patient is pregnant or lactating
* The patient has had prior breast radiation to the ipsilateral breast
* The patient has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes
* The patient has recevied a Feraheme (ferumoxytol) injection within the past 6 months
* The patient has intolerance or hypersensitivity to iron or dextran compounds or to Magtrace
* The patient has iron overload disease
* The patient has discoloration on the breast (such as tattoo, birthmark, tanning, rash etc.), that in the Investigator's opinion, could impact the clinical trial results, specifically the assessment of any skin discoloration, or plans to have a tattoo on the breast post-operatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects considered for enrollment will be at least 18 years old at the time of consent, and: a) due to undergo planned breast conserving surgery (for example lumpectomy or partial mastectomy) and SLNB with Magtrace b) meet all other inclusion and no exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of Magtrace-related skin discoloration as a proportion of patients receiving Magtrace, overall and by sub-sample | post-op to 24 month follow-up
  Frequency of Magtrace-related skin discoloration as a proportion of patients receiving Magtrace, overall and by sub-sample

SECONDARY OUTCOMES:
Change in BREAST-Q score from post-operative visit through to resolution of skin discoloration or through 24 months, whichever is earlier, in the subgroup of patients with discoloration. 7 core scales will be used. | Baseline to 24 month follow-up
Change in BREAST-Q score from pre-operative visit to post-operative visit in patients with and without skin discoloration at the post-op follow-up visit. | Pre-op to Post-Op
Duration of discoloration over time post-op to resolution of discoloration or 24 month follow-up | Post-op to 24 month follow-up
Intensity of discoloration (absolute color and contrast to normal breast color) over time post-op to resolution of discoloration or 24 month follow-up | Post-Op to 24 month follow-up
Severity of discoloration over time post-op to resolution of discoloration or 24 month follow-up as assessed by height and width measurement | Post-Op to 24 month follow-up
Rates of device-related adverse events and serious device-related adverse events | Baseline to 24 month follow-up
Number of identified SLNs per patient | Surgery
  Number of identified SLNs per patient
Number of non-Magtrace marked nodes per patient removed (clinically suspicious) | Surgery
  Number of non-Magtrace marked nodes per patient removed (clinically suspicious).
Nodal malignancy rate | Surgery
  Nodal malignancy rate

OTHER OUTCOMES:
Overall SLN detection rate (proportion of patients with successful SLN detection using Magtrace) | Surgery
  Overall Sentinel Lymph Node detection rate - proportion of patients with successful SLN detection using Magtrace

CONTACTS AND LOCATIONS:
Locations (1):
- VCU Massey Comprehensive Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No